CLINICAL TRIAL: NCT05667402
Title: Clinical Study of TBF Regimen in Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Central Nervous System Leukemia
Brief Title: Clinical Study of TBF Regimen in Allo-HSCT in Patients With CNS Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-307
Record Dates: First submitted 2022-10-27; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-10

CONDITIONS: Central Nervous System Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBF group (Experimental): The subjects receive TBF conditioning regimen.
  Interventions: Drug: TBF regimen
- Modified BuCY2 group (Active Comparator): The subjects receive modified BuCY2 conditioning regimen.
  Interventions: Drug: modified BuCY2 regimen

INTERVENTIONS:
Drug: TBF regimen — The subjects receive TBF conditioning regimen (Thiotepa, Busulfan, Fludarabine) before allo-HSCT.
  Other Names: Conditioning treatment with TBF regimen
  Arms: TBF group
Drug: modified BuCY2 regimen — The subjects receive modified BuCY2 conditioning regimen (Busulfan, Cytarabine, ATG, Cyclophosphamide, CCNU) before allo-HSCT.
  Other Names: Conditioning treatment with modified BuCY2 regimen
  Arms: Modified BuCY2 group

SUMMARY:
Central nervous system (CNS) leukemia is a poor prognostic factor for allogeneic hematopoietic stem cell transplantation (allo-HSCT). Thiotepa can penetrate the blood-brain barrier and has immunosuppressive effects and similar effects to irradiation in allo-HSCT. This project aims to investigate whether the TBF regimen is superior to the traditional modified BuCY2 regimen to improve the long-term survival of the CNS leukemia patients.

DETAILED DESCRIPTION:
Central nervous system (CNS) leukemia is a common extramedullary leukemia and a poor prognostic factor for allogeneic hematopoietic stem cell transplantation (allo-HSCT). There is a blood-brain barrier (BBB) in the CNS. The treatment effect of CNS leukemia is seriously limited by the low penetration of conventional chemotherapy drugs into cerebrospinal fluid. Thiotepa can penetrate the BBB and has immunosuppressive effect and myeloablative effect similar to irradiation in transplantation. Therefore, it is speculated that cestipide has certain advantages as a conditioning regimen in transplantation for CNS leukemia. This project aims to investigate whether the TBF regimen is superior to the traditional modified BuCY2 regimen to improve the long-term survival of the CNS leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with central nervous system leukemia by MICM meet one of the following conditions: corresponding symptoms and signs of central nervous system involvement; cerebrospinal fluid pressure increased by 200 mm water column; the white blood cell count in cerebrospinal fluid was 0.01×10^9/L; cerebrospinal fluid protein qualitative test was positive or protein quantification was 45 mg/dL; leukemic cells can be found in the cerebrospinal fluid; cranial imaging suggested central involvement.
* Aged 14-60 years, male or female.
* KPS score: ≥80.
* Signed the informed consent.

Exclusion Criteria:

* Patients intending to receive autologous hematopoietic stem cell transplantation.
* Patients with transplantation contraindications.
* Those who refuse to sign the informed consent form.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of central nervous system (CNS) leukemia | From date of the treatment with the conditioning regimen until CNS leukemia relapse, the end of follow-up or the date of death from any cause, whichever came first, assessed up to 36 months.
  The proportion of patients with recurrent central nervous system leukemia in the total enrolled population

SECONDARY OUTCOMES:
Hematopoietic implantation rate | From date of the treatment with the conditioning regimen until hematopoietic implantation, assessed up to 100 days..
  Hematopoiesis was achieved within 100 days after allo-HSCT
NRM | From date of allo-HSCT until the date of death from any cause or the end of follow-up, whichever came first, assessed up to 36 months.
  non-recurrence mortality
OS | From date of the treatment with the conditioning regimen until the end of follow-up or the date of death from any cause, whichever came first, assessed up to 36 months.
  overall survival
PFS | From date of the treatment with the conditioning regimen until leukemia progression, the end of follow-up or the date of death from any cause, whichever came first, assessed up to 36 months.
  progression-free survival
AEs | From date of the treatment with the conditioning regimen until the occurrence of adverse effects, the end of follow-up or the date of death from any cause, whichever came first, assessed up to 36 months.
  adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, MD, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China